CLINICAL TRIAL: NCT00793260
Title: Deep Dive Randomized Control Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Health Dialog (Industry)
Collaborators: Health Net California (Unknown); Highmark Blue Cross Blue Shield (Unknown)
Responsible Party: David E. Wennberg, MD, MPH / Chief Science & Products Officer, Health Dialog Analytic Solutions, Inc
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: DeepDive
Record Dates: First submitted 2008-11-17; First posted 2008-11-19 (Estimated); Last update posted 2008-11-19 (Estimated); Status verified 2008-11

CONDITIONS: Chronic Disease; Arthritis; Uterine Diseases; Spinal Diseases; Preventive Health Services
MeSH Terms: conditions — Chronic Disease; Arthritis; Uterine Diseases; Spinal Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual Support Group (Active Comparator): Predictive models in the Usual-Support Group were aimed at identifying individuals through medical claims and administrative data (such as hospitalization notification). The output of the predictive models is a rank-ordered, or stratified, list of individuals who have support needs. These lists were then used to generate outbound mail, interactive voice response (IVR) calls or calls by health coaches.
  Interventions: Behavioral: Usual-Support
- Enhanced Support Group (Experimental): The Enhanced-Support Group intervention used more sophisticated predictive models, more extensive outreach to engage individuals, and provided tighter feedback loops to inform the care support process.
  Interventions: Behavioral: Enhanced Support

INTERVENTIONS:
Behavioral: Enhanced Support — The Enhanced-Support Group program used lower risk thresholds for targeted outreach of individuals with chronic illness and for those likely to face discrete surgical interventions. Individuals at high financial risk but without one of the five chronic conditions were included in the Enhanced-Support Group.
  The Enhanced-Support Group received up to five initial reach attempts while the Usual-Support Group received up to three attempts.
  The Enhanced-Support Group used a 'tight loop' management structure including detailed, timely coach level feedback reports on efficiency and effectiveness.
  Arms: Enhanced Support Group
Behavioral: Usual-Support — Predictive models in the Usual-Support Group were aimed at identifying individuals through medical claims and administrative data (such as hospitalization notification). The output of the predictive models is a rank-ordered, or stratified, list of individuals who have support needs. These lists were then used to generate outbound mail, interactive voice response (IVR) calls or calls by health coaches.
  Arms: Usual Support Group

SUMMARY:
Compare two care management support program models on medical costs and utilization.

ELIGIBILITY:
Inclusion Criteria:

* All employees, dependents and retirees in one of seven large employer groups, including a state university system, a state employee group, two manufacturing companies, a natural resource extraction company, a public educational service agency, and a nonprofit multiple employer association for independent colleges were eligible for inclusion.

Exclusion Criteria:

* no financial information was available from their facility and professional claims;
* they were in an employer sub-group ineligible for care support services;
* they asked not be to contacted or were deceased;
* gender information was missing from their eligibility files;
* their claims data from the year prior to the start of the study indicated diagnoses of HIV, AIDS, end-stage renal disease (ESRD), organ transplants, or necrotizing fasciitis (intended to improve the likelihood of a balanced distribution of costs and conditions); OR
* they were in an employer sub-group with less than four months of enrollment prior to the study start date (resulting in too little information for stratification).

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 174120 (Actual)
Dates: Start 2006-07; Primary Completion 2007-06 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure was total medical costs (capped at $200,000 per individual per year) and pharmacy costs.

SECONDARY OUTCOMES:
Secondary measures included utilization of selected services.

CONTACTS AND LOCATIONS:
Overall Officials: David E Wennberg, MD, MPH, Principal Investigator — Health Dialog
Locations (1):
- Health Dialog Analytic Solutions, Inc, Portland, Maine, United States

REFERENCES:
- [Derived] Wennberg DE, Marr A, Lang L, O'Malley S, Bennett G. A randomized trial of a telephone care-management strategy. N Engl J Med. 2010 Sep 23;363(13):1245-55. doi: 10.1056/NEJMsa0902321. PMID 20860506